CLINICAL TRIAL: NCT05234515
Title: Prospective Bacteriology of sUrGical Site INfection Following Surgery for Intestinal Failure
Brief Title: Bacteriology of sUrGical Site INfection Following Surgery for Intestinal Failure
Acronym: BUGS-IN-IF
Status: Completed | Type: Observational
Sponsor: London North West Healthcare NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: RD21/049; 301274 (Other: IRAS)
Record Dates: First submitted 2021-10-28; First posted 2022-02-10 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2022-10

CONDITIONS: Surgical Wound Infection; Surgical Site Infection; Bacteria Infection Mechanism; Intestinal Disease; Intestinal Fistula
MeSH Terms: conditions — Surgical Wound Infection; Intestinal Diseases; Intestinal Fistula | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Bacterial culture
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with intestinal failure or an enterocutaneous fistula undergoing elective surgery.: Adult patients with a diagnosis of intestinal failure (IF) or an enterocutaneous fistula (ECF) undergoing planned surgery in our unit.
  Interventions: Diagnostic Test: Microbiology swab; Other: Questionnaire

INTERVENTIONS:
Diagnostic Test: Microbiology swab — Patients will have swabs taken from the nose, mouth, umbilical skin, groin skin, fistula(e), stoma(s) and vascular access device prior to surgery. Patients will be followed for 90 days postoperatively for surgical site infection (SSI) as defined by the centre for disease control (CDC) criteria 2021. Patients who develop an SSI will have both preoperative and postoperative samples sent for genome sequencing.
Other: Questionnaire — Patients will complete baseline preoperative questionnaires which will be repeated at 30 days and 90 days. These will evaluate generic and wound specific quality of life as well as decision conflict/decision regret.

SUMMARY:
This is a prospective observational study of patients undergoing planned surgery for intestinal failure. The aims of the study are:

* To prospectively characterise preoperative bacterial populations amongst patients undergoing surgery for intestinal failure
* To examine the relationship between preoperative bacteriology and surgical site infection (SSI) in this patient group
* To investigate the effect of surgery and surgical site infection on generic and wound specific quality of life measures

ELIGIBILITY:
Inclusion Criteria:

* Adults aged >18 year
* Diagnosis of intestinal failure or enterocutaneous fistula
* Undergoing elective surgery within St Mark's hospital IF unit

Exclusion Criteria:

* Unable or unwilling to provide informed consent
* Pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited from the intestinal failure unit at St Mark's hospital, London North West University Healthcare NHS Trust.
Sampling Method: Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2022-01-14 (Actual); Primary Completion 2022-10-30 (Actual); Study Completion 2023-02-20 (Actual)

PRIMARY OUTCOMES:
Clinical Surgical Site Infection (SSI) | 0-90 days
  Classified as either superficial, deep or organ space as defined by the centre for disease control (CDC) classification 2021
Microbiological | 0-90 days
  Preoperative colonisation species, Organisms cultured from SSI, Correlation to preoperative samples
Change in Generic Quality of Life Score | Baseline - 90 days
  Generic health scores quantified by the validated EuroQoL 5 dimension, 5 level questionnaire (EQ5D-5L) at baseline, 30 and 90 days. (Minimum score 5, Maximum score 25)
Change in Wound Specific Quality of Life Score | Baseline - 90 days
  Quantified by the Wound-QoL questionnaire, a validated 17 item scale at baseline, 30 and 90 days (Minimum score 0, Maximum score 68)
Decision conflict | Day 0
  Preoperative decision conflict scores quantified by decision conflict scale (DCS), a validated 16 point scale (Minimum score 0, Maximum score 64)
Change in Decision Regret | 30 and 90 days
  Postoperative decision regret scores quantified by the decision regret scale (DRS) a validated 5 item questionnaire, at 30 and 90 days. (Minimum score 5, Maximum score 25)

SECONDARY OUTCOMES:
Length of stay | from day of surgery (day 0)
  Duration of index hospital admission, measured in days
Complications | 90 days
  Classified using the Clavien-Dindo classification(I-V)
Abdominal wound healing | 90 days
  Classified as either 'completely healed' OR 'incompletely healed'

CONTACTS AND LOCATIONS:
Overall Officials: Carolynne F Vaizey, Principal Investigator — St Marks Hospital & Academic Institute
Locations (1):
- St Marks Hospital, Harrow, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared. Summary findings will be disseminated to other health care workers and patient groups at conference where the work will be presented. The data will be submitted to a peer-reviewed medical journal for publication. Internal reports will update on the progress of the work. The data will be under the ownership of London north west university healthcares trust (LNWUHT). The PhD student involved, and their team will have rights to publish the data. Patient participants will be notified of publications and asked if they would like to receive copies following the study period.